CLINICAL TRIAL: NCT00220233
Title: Add-on Study of Olmesartan Medoxomil in Patients With Moderate to Severe Hypertension Not Achieving Target Blood Pressure on Amlodipine 5 mg Alone
Brief Title: Olmesartan as an add-on to Amlodipine in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS8663-A-E303
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2007-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Amlodipine; Hydrochlorothiazide

INTERVENTIONS:
Drug: olmesartan medoxomil
Drug: amlodipine
Drug: hydrochlorothiazide

SUMMARY:
This study is to test the efficacy and safety of the combination of olmesartan and amlodipine in hypertensive patients whose blood pressure is not adequately controlled with amlodipine alone

ELIGIBILITY:
Inclusion Criteria:

* Without antihypertensive pre-treatment mean seated BP greater than 160/100 mmHg
* Pre-treatment with amlodipine 5 or 10 mg: mean seated BP greater than or equal to 140/90 mmHg

Exclusion Criteria:

* Secondary hypertension
* Any serious disorder which may limit the ability to evaluate the efficacy or safety of the test drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632
Dates: Start 2005-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean change in trough seated diastolic blood pressure

SECONDARY OUTCOMES:
Mean change in trough seated systolic BP
Mean change in daytime, nighttime and 24 hour ambulatory blood pressure
Percent of patients achieving target blood pressure goal
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brommer, MD, Principal Investigator
Locations (5):
- Germany (5):
  - Leipzig
  - Sinsheim
  - Tann
  - Weinheim
  - Wiesbaden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/